CLINICAL TRIAL: NCT05833529
Title: Virtual Reality Cue Exposure Therapy for Cocaine Craving: an Innovative Cognitive and Behavioral Psychotherapy for Cocaine Use Disorder (Psychothérapie Innovante COmportementale et Cognitive Pour le Trouble d'Usage de Cocaïne; PICOC)
Brief Title: Innovative Cognitive and Behavioral Psychotherapy for Cocaine Use Disorder
Acronym: PICOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Lehoux (Other)
Collaborators: Laboratoire de Psychologie des Cognitions (Strasbourg University, France) (Unknown); ICube Laboratory - Team IGG (Strasbourg University, France) (Unknown); Hospital Center of Saint-Esprit (Martinique) (Unknown); National Cancer Institute, France (Other Government); French Institute for Public Health Research (IReSP) (Unknown); GIRCI SOHO (Other)
Responsible Party: Sponsor-Investigator, Thomas Lehoux, Ph.D. Candidate, University Hospital Center of Martinique
Organization: University Hospital Center of Martinique (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22_RIPH2-18; 2022-A02440-43 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-03-27; First posted 2023-04-27 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine; Virtual Reality Cue Exposure Therapy; Craving; Cognitive and Behavioral Therapy; Cue Exposure Therapy; Memory Focused Cognitive Therapy; Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRCET for Cocaine Craving then MFCT (Experimental): 3 weeks treatment consisting of 10 meetings of Virtual Reality Cue Exposure Therapy (VRCET) for cocaine craving, followed by 5 meetings of Memory Focused Cognitive Therapy (MFCT). All meetings will last 90 minutes. VRCET meetings will take place in a 2 weeks period (weeks 1 and 2) at a daily frequency from monday to friday included. MFCT meetings will take place in the 1 week period following VRCET (week 3) at a daily frequency from monday to friday included.
  Interventions: Behavioral: Virtual Reality Cue Exposure (VRCE) Therapy for Cocaine Craving - 2 weeks; Other: Memory Focused Cognitive Therapy (MFCT) - 1 week
- PCET for Cocaine Craving (Active Comparator): 3 weeks treatment consisting of 15 meetings of Picture-based Cue Exposure Therapy (PCET) for cocaine craving. All meetings will last 90 minutes. PCET meetings will take place in a 3 weeks period (weeks 1 to week 3) at a daily frequency from monday to friday included.
  Interventions: Behavioral: Pictures-based Cue Exposure (PCE) Therapy for Cocaine Craving - 3 weeks

INTERVENTIONS:
Behavioral: Virtual Reality Cue Exposure (VRCE) Therapy for Cocaine Craving - 2 weeks — 40 10 mins VRCEs for cocaine craving (desensitization to only cocaine craving cues; no others interventions). 4 VRCE and 2 different VRCE situations by meeting. Same VRCE situations spaced intra (30 mins) and inter meetings (48 hrs). 5 standard VRCE situations (appearance and dialogues adapted to Martinique field) varying from "only peers cocaine use talk" to "peers and participant prepare and use cocaine" and ranging from the lowest to the highest participant related cocaine craving level. Situation switch to another when its initial cocaine craving level has decreased to its half for 5 continuous VRCE mins (must be ≤ 3/10; 0 = none; 10 = very high). Meetings end with relaxation/relapse prevention in any case of distress still over convenient levels. VRCE use Meta Quest 2, are visuo-auditively immersive (360°; 1st person), interactive (using virtual objects), semi-stationnary (360°-rotating stool and teleportation system). Participant skin color and cocaine using mode individualized.
  Arms: VRCET for Cocaine Craving then MFCT
Other: Memory Focused Cognitive Therapy (MFCT) - 1 week — In accordance with the "Memory Focused Cognitive Therapy for Cocaine Use Disorder" Therapist Guide (Marsden and Goetz, 2018), MFCT meetings will consist in 5 sequential components: Cognitive case conceptualisation of cocaine use disorder maintaining processes to inform a treatment plan; Education about cocaine's cognitive and physical effects; Cocaine related cue-induction to elicit images and affective responses; Memory reconsolidation procedures; Standard CBT techniques (e.g. behavioural experiments of cocaine-related expectancies and skills for adaptive emotion regulation).
  Arms: VRCET for Cocaine Craving then MFCT
Behavioral: Pictures-based Cue Exposure (PCE) Therapy for Cocaine Craving - 3 weeks — 60 x 10 mins PCE (desensitization to only cocaine craving cues; no others interventions). A standard audio of VRE songs is played in PCE. 4 PCE and 2 different PCE situations by meeting. Same PCE situations spaced intra (30 mins) and inter meetings (48 hrs). 5 standard PCE situations (appearance and dialogues adapted to Martinique field) varying from "only peers cocaine use talk" to "peers and participant prepare and use cocaine" and ranging from the lowest to the highest participant related cocaine craving level. Situation switch to another when its initial cocaine craving level has decreased to its half for 5 continuous PCE mins (must be ≤ 3/10; 0 = none; 10 = very high). Meetings end with relaxation/relapse prevention if any distress over convenient levels. PCE use a laptop standard PowerPoint slide show (2D pictures from VRCE; non-spatialized audio from laptop speakers), are non-interactive (seated on a stool). Participant skin color and cocaine using mode individualized.
  Arms: PCET for Cocaine Craving

SUMMARY:
Cocaine is the 2nd most used illicit substance in Europe and its use implies numerous health complications as well as an annual social cost of 8.7 G d'€. Classical (picture, video, audio, imagery based or in vivo) cue exposure therapy for substance craving (CET), i.e. the irrepressible and non-voluntary desire to use the substance, failed to prove efficacious in treating substance use disorder. Virtual reality cue exposure therapy for substance craving (VRCET), is more immersive, realistic and controllable, and is suggested as being a more efficacious intervention in reducing craving as compared to classical CET.

So far it's still not known, thus the secondary aim of the present randomized and clinical trial is to investigate, whether virtual reality cue exposure is more efficacious, as compared to classical cue exposure, in both eliciting and reducing cocaine craving in a clinical context of CET for cocaine craving. The main study aim to is to investigate whether a VRCET for cocaine craving based cognitivo-behavioral therapy (i.e. VRCET followed by memory focused cognitive therapy) is more efficacious than a behavioural therapy (i.e. classical exposure therapy to craving) in reducing cocaine craving.

To do so, 54 voluntary residential patients in treatment for cocaine use disorder will be recruited from the Universitary Hospital Center of Martinique (CHUM, Martinique, France) and Saint-Esprit Hospital Center (CHSE, Martinique, France) and randomly allocated in either a 3 weeks individual experimental treatment (10 meetings of VRET for cocaine craving followed by 5 meetings of memory focused cognitive therapy) or a 3 weeks individual control treatment (15 meetings of pictures based exposure therapy for cocaine craving). Self-reported measures of retrospective (last 14 days) and in virtuo exposure cocaine craving will be collected at the beginning, after 10 days, after 15 days of treatment and 1 month post. Others secondary subjective, urinary and physiological cocaine use related measures will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age greater than or equal to 18),
* Present the diagnostic criteria for a cocaine use disorder (DSM-5; SCID 5-CV),
* Be voluntarily hospitalized and engaged in a residential standard treatment for cocaine use disorder at the Universitary Hospital of Martinique or at the Hospital Centre of Saint-Esprit in Martinique,
* Present a motivation of "action" or "maintenance" of cocaine use cessation (University of Rhode Island Change Assessment Scale),
* Have been informed of the research,
* Have given free, informed and express consent,
* Be affiliated to a social security scheme.

Exclusion Criteria:

* Present the diagnostic criteria (MINI 5.0.0.; DSM-IV):

  * Current high suicide risk episode,
  * Current psychotic syndrome,
  * Current mania or hypomania episode,
  * Current post-traumatic stress
* Present significant symptoms of cyberkinetosis in virtual reality exposure (SP-IE),
* Present another current medical condition at risk of danger or inability to comply with the protocol (e.g. heart problems, blindness or deafness,...),
* Be placed under legal safeguard, guardianship or curatorship,
* Patient who refused to participate in the study,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cocaine Craving Intensity (in Virtual Reality Cue Exposure for Cocaine Craving) at the End of Treatment | Right before treatment and at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3)
  Self-reported cocaine craving intensity in virtuo exposure to cocaine craving according to the Craving Expérience Questionnaire (french version; CEQ-F "Envie la Plus Forte" total score; Ceschi et Pictet, 2018). CEQ-F "Envie la Plus Forte" total score varies from 11 to 111 (higher score suggesting higher craving intensity). CEQ-F "Envie la Plus Forte" is administrated immediatly after a standard 5 mins virtual reality cue exposure for cocaine craving and focuses on the strongest cocaine craving felt during the exposure. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Change from Baseline Cocaine Craving Frequency (Last 14 Days) at the End of Treatment | Right before treatment and at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3)
  Self-reported retrospective cocaine craving frequency in the last 14 days according to the Craving Expérience Questionnaire (french version; CEQ-F "A Quelle Fréquence" total score; Ceschi et Pictet, 2018). CEQ-F "A Quelle Fréquence" total score varies from 11 to 111 (higher score suggesting higher craving frequency). CEQ-F "A Quelle Fréquence" focuses on the frequence of cocaine craving in the last 14 days.

SECONDARY OUTCOMES:
Cocaine Craving Intensity (in Virtual Reality Cue Exposure for Cocaine Craving) | Right before treatment; at the end of each VR or pictures-based exposures during VRCET and PCET; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported cocaine craving intensity in virtuo exposure to cocaine craving according to the Craving Expérience Questionnaire (french version; CEQ-F "Envie la Plus Forte" total score; Ceschi et Pictet, 2018). CEQ-F "Envie la Plus Forte" total score varies from 11 to 111 (higher score suggesting higher craving intensity). CEQ-F "Envie la Plus Forte" is administrated immediatly after a standard 5 mins virtual reality cue exposure for cocaine craving and focuses on the strongest cocaine craving felt during the exposure. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Cocaine Craving Frequency (Last 14 Days) | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported retrospective cocaine craving frequency in the last 14 days according to the Craving Expérience Questionnaire (french version; CEQ-F "A Quelle Fréquence" total score; Ceschi et Pictet, 2018). CEQ-F "A Quelle Fréquence" total score varies from 11 to 111 (higher score suggesting higher craving frequency). CEQ-F "A Quelle Fréquence" focuses on the frequence of cocaine craving in the last 14 days.
Cocaine Craving Occurence, Imagery and Intrusiveness Frequency (Last 14 Days) | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported retrospective cocaine craving occurence, imagery and intrusiveness frequency in the last 14 days according to the Craving Expérience Questionnaire (french version; CEQ-F "A Quelle Fréquence" subscales total scores; Ceschi et Pictet, 2018). CEQ-F "A Quelle Fréquence" higher subscales total scores suggesting higher frequencies).
Cocaine Craving Occurence, Imagery and Intrusiveness Intensity (in Virtual Reality Cue Exposure for Cocaine Craving) | Right before treatment; at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported cocaine craving occurence, imagery and intrusiveness intensity in virtuo exposure to cocaine craving according to the Craving Expérience Questionnaire (french version; CEQ-F "Envie la Plus Forte" subscales total scores; Ceschi et Pictet, 2018). CEQ-F "Envie la Plus Forte" higher subscales total scores suggesting higher intensities). CEQ-F "Envie la Plus Forte" subscales are administrated immediatly after a standard 5 mins virtual reality cue exposure for cocaine craving and focuses on the strongest cocaine craving felt during the exposure. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Negatives and Positive Emotional States (in Virtual Reality Cue Exposure for Cocaine Craving) | Right before treatment; at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported intensity of negative and positive emotional states in virtuo exposure to cocaine craving according to the Brief Mood Introspection Scale (french version; BMIS negative and positive subscales total scores; Dalle et al., 2003). BMIS higher subscales total scores suggesting higher intensities). BMIS subscales are administrated immediatly after a standard 5 mins virtual reality cue exposure for cocaine craving. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Self-Efficacy to Cope with Cocaine Craving without Using (in Virtual Reality Cue Exposure for Cocaine Craving) | Right before treatment; at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported efficacy to cope with cocaine craving in virtuo exposure to cocaine craving according to the Drug Taking Confidence Questionnaire 8D (french version; DTCQ-8D total score; Sklar et al., 1999). DTCQ-8D higher total score suggesting higher self-efficacy). DTCQ-8D is administrated immediatly after a standard 5 mins virtual reality cue exposure for cocaine craving. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Blood Volume Pulse and Skin Temperature (in Virtual Reality Cue Exposure for Cocaine Craving) | Right before treatment; at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Blood volume pulse and skin temperature in virtuo exposure to cocaine craving according to PLUX Biosignals medically certificated devices (# ISO-13485; https://www.pluxbiosignals.com/pages/about). Blood volume pulse and skin temperature are recorded during a standard 5 mins virtual reality cue exposure for cocaine craving. The virtual reality cue exposure environment is different from the one to which participants were exposed during treatment, in contrary to VR settings which are similar.
Spatial Presence, Sense of Reality and Cybersickness related to Cue Exposure Environments for Cocaine Craving | Before treatment; during treatment phase at each new cue exposure situation for cocaine craving experienced
  Self-reported spatial presence, sense of reality and cybersickness related to cue exposure environments according to the Spatial Presence for Immersive Environments (french version; SP-IE subscales total scores; Khenak et al., 2019). SP-IE subscales "sense of spatial presence", "the affordance of the environment", "the user's enjoyment", "the user's attention allocation to the task", "the sense of reality attributed to the environment", "the social embodiment with avatars", and "the possible negative effects of the environment (cybersickness)" are administrated immediatly after each new cue exposure environment experienced.
Ecological Validity related to Cue Exposure Environments for Cocaine Craving | Before treatment; during treatment phase at each new cue exposure situation for cocaine craving experienced
  Self-reported ecological validity related to cue exposure environments according to the Independant Television Commission - Sense Of Presence Inventory (french version; ITC-SOPI subscale total score; I2 Media Research Ltd, 2004; Independent Television Commission, 2000). The ITC-SOPI subscale "Ecological Validity/Naturalness" is administrated immediatly after each new cue exposure environment experienced.
Propensity to Cocaine Relapse (Next 2 Months) | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self-reported propensity to cocaine relapse in the next 2 months according to the Advance WArning of RElapse scale (french translated version; AWARE total score; Miller and Harris, 2000; Kelly and al., 2011).
Dysfonctional Beliefs related to Cocaine Use | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Identification level to dysfunctional beliefs to cocaine use according to the Questionnaire of Core Beliefs related to Drug Use and Craving (french translated version; QBDU - Belief related to Addiction subscale total score; Martinez-Gonzalez et al., 2018).
Abstinence from Cocaine Use (Retrospective) | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self reported retrospective measure of abstinence from cocaine use in the last 14 days according to the Timeline Followback (french translated version; TLFB total score; Sobell and Sobell, 1992; Mapi Institute, 2012).
Abstinence from Cocaine Use (Urine Drug Testing) | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Medical certified device of urinary drug testing measure of cocaine use in the last 7 days (Universitary Hospital Center of Martinique CSAPA, 2023).
Emotions Dysregulation | Right before treatment; at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3); 1 month post treatment (week 7)
  Self reported questionnaire measure of emotion dysregulation according to the Difficulties in Emotion Regulation Scale (french version; DERS total score; Côté et al., 2013).
Client Satisfaction related to the Therapy | at the end of "VRCET" and "PCET" 2 weeks (week 2); at the end of "VRCET then MFCT" and "PCET" (end of treatment; week 3)
  Self reported questionnaire measure of client satisfaction related to the therapy according to the Client Satisfaction Questionnaire 8 (french version; CSQ 8 total score; Sabourin and al., 1989; Attkisson, 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme LACOSTE, MD, Principal Investigator — CHU of Martinique; Thomas LEHOUX, Ph.D. Candidate, Study Director — Laboratoire de Psychologie des Cognitions (Strasbourg University, France)
Locations (2):
- Martinique (2):
  - University Hospital Center of Martinique, Fort-de-France
  - Hospital Center of Saint-Esprit (Martinique), Saint-Esprit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conklin CA, Tiffany ST. Applying extinction research and theory to cue-exposure addiction treatments. Addiction. 2002 Feb;97(2):155-67. doi: 10.1046/j.1360-0443.2002.00014.x. PMID 11860387
- [Background] Lee JH, Ku J, Kim K, Kim B, Kim IY, Yang BH, Kim SH, Wiederhold BK, Wiederhold MD, Park DW, Lim Y, Kim SI. Experimental application of virtual reality for nicotine craving through cue exposure. Cyberpsychol Behav. 2003 Jun;6(3):275-80. doi: 10.1089/109493103322011560. PMID 12855083
- [Background] Marsden J, Goetz C, Meynen T, Mitcheson L, Stillwell G, Eastwood B, Strang J, Grey N. Memory-Focused Cognitive Therapy for Cocaine Use Disorder: Theory, Procedures and Preliminary Evidence From an External Pilot Randomised Controlled Trial. EBioMedicine. 2018 Mar;29:177-189. doi: 10.1016/j.ebiom.2018.01.039. Epub 2018 Feb 2. PMID 29478874
- [Background] Hone-Blanchet A, Wensing T, Fecteau S. The use of virtual reality in craving assessment and cue-exposure therapy in substance use disorders. Front Hum Neurosci. 2014 Oct 17;8:844. doi: 10.3389/fnhum.2014.00844. eCollection 2014. PMID 25368571
- [Background] Saladin ME, Brady KT, Graap K, Rothbaum BO. A preliminary report on the use of virtual reality technology to elicit craving and cue reactivity in cocaine dependent individuals. Addict Behav. 2006 Oct;31(10):1881-94. doi: 10.1016/j.addbeh.2006.01.004. Epub 2006 Mar 3. PMID 16516397
- [Derived] Lehoux T, Capobianco A, Lacoste J, Rollier S, Mopsus Y, Melgire M, Lecuyer F, Gervilla M, Weiner L. Virtual reality cue-exposure therapy in reducing cocaine craving: the Promoting Innovative COgnitive behavioral therapy for Cocaine use disorder (PICOC) study protocol for a randomized controlled trial. Trials. 2024 Jun 27;25(1):421. doi: 10.1186/s13063-024-08275-7. PMID 38937824